CLINICAL TRIAL: NCT07226661
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of SPN-821 as an Adjunctive Therapy in Adults With Major Depressive Disorder
Brief Title: Double-blind, Placebo-controlled Study in Adults With Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 821P203
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPN-821 2400 mg (Experimental): Three 800 mg oral tablets administered twice a week adjunctive to current antidepressant
  Interventions: Drug: SPN-821 2400 mg
- Placebo (Placebo Comparator): Three oral tablets administered twice a week adjunctive to current antidepressant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-821 2400 mg — SPN-821 is a novel, orally bioavailable, selective, direct enhancer of mTORC1 cellular signaling
  Arms: SPN-821 2400 mg
Drug: Placebo — Matched placebo oral tablets
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of SPN-821 in adults with major depressive disorder

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of SPN-821 administered twice a week as adjunctive therapy to an approved antidepressant therapy in adult participants with MDD. The study includes a 2-week Screening Period, a 4-week Double blind Treatment Period, and a Safety Follow-up phone call one week after the completion of the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of MDD according to the DSM-5 for either single or recurrent MDE without psychotic features confirmed by the MINI
* Duration of current MDE of at least 8 weeks
* MADRS total score of ≥ 24 at the Screening Visit and Day 1 Visit
* CGI-S score of ≥ 4 (moderately ill or worse) at the Screening Visit and Day 1 Visit
* Stable, therapeutic dose of one of the following protocol-approved ADTs as a monotherapy for ≥ 8 weeks before the Screening Visit and ≥ 10 weeks at the Day 1 Visit. Additionally, inadequate response to the current ADT (less than 50% improvement in depressive symptoms) as confirmed by the ATRQ Investigator administered.

Exclusion Criteria:

* MADRS total score change of ≥ 25% from the Screening Visit to Day 1 Visit
* History of treatment resistant depression (TRD) defined as 3 or more failed ADTs of adequate dose (per ATRQ) and duration (at least 8 weeks) for the current MDE
* History of alcohol or substance use disorder according to DSM-5 criteria 6 months before the Screening Visit
* Evidence of significant risk for suicidal behavior during participation in the study in the Investigator's opinion
* Lifetime diagnosis of any psychotic disorder including MDD with psychosis, MDD with mixed features, bipolar I/II disorder, bipolar depression, schizophrenia, posttraumatic stress disorder, autism spectrum disorder, or any personality disorder or intellectual disability that would affect the ability of the participant to enroll in the study
* Diagnosis less then 12 months before screening of severe obsessive-compulsive disorder, acute stress disorder, panic disorder, eating disorders, or any other psychiatric condition that has been the primary focus of treatment, or diagnosis of generalized anxiety disorder less then 6 months before screening.
* History of cardiovascular, respiratory, gastrointestinal, renal, hepatic, and hematologic disorders, or other medical disorders that could impose undue risk or compromise the study in the Investigator's opinion
* Clinically significant abnormal result prior to Day 1 Visit per Investigator's judgment or abnormal renal function.
* Requires treatment with a medication or other substance that is prohibited by the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Day 29 in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score. | 4 weeks
  MADRS is a 10-item scale (Reported sadness, Apparent sadness, Inner tension, Reduced sleep, Reduced appetite, Concentration difficulties, Lassitude, Inability to feel, Pessimist thoughts, and Suicidal thoughts) where each item is scored from 0 to 6. The total score is the sum of the 10 items ranging from 0 to 60 where higher scores indicate more severe depression, and lower scores are better outcomes.

SECONDARY OUTCOMES:
Change From Baseline to Day 29 in the Clinical Global Impression - Severity of Illness Score (CGI-S). | 4 weeks
  CGI-S is a single-item clinician rating of the clinician's assessment of the severity of symptoms in relation to the clinician's total experience with patients with that condition. The CGI-I is rated on a 7-point scale from 1 to 7, where 1 = "normal not at all ill" and 7 = "among the most extremely ill patients". Successful therapy is indicated by a lower overall score.

CONTACTS AND LOCATIONS:
Locations (1):
- Collaborative Neuroscience Network, Garden Grove, California, United States

IPD SHARING:
Plan to Share IPD: No